CLINICAL TRIAL: NCT00162981
Title: Safety and Efficacy of Clobazam in Subjects With Lennox-Gastaut Syndrome
Brief Title: Clobazam in Subjects With Lennox-Gastaut Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13108A; OV1002 (Other: Former study ID)
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2012-02-09 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2012-01

CONDITIONS: Epilepsy; Epilepsy, Generalized; Seizures
MeSH Terms: conditions — Epilepsy; Epilepsy, Generalized; Seizures | interventions — Clobazam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clobazam Low Dose (Experimental)
  Interventions: Drug: Clobazam Low Dose
- Clobazam High Dose (Experimental)
  Interventions: Drug: Clobazam High Dose

INTERVENTIONS:
Drug: Clobazam Low Dose — 5 to 10 mg/day with doses in the morning and at bedtime; orally
  Other Names: Onfi™
  Arms: Clobazam Low Dose
Drug: Clobazam High Dose — 5 to 40 mg/day with doses in the morning and at bedtime; orally
  Other Names: Onfi™
  Arms: Clobazam High Dose

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of clobazam as adjunctive therapy in the treatment of seizures which lead to drop attacks (drop seizures) in subjects 2 to 30 years of age with Lennox-Gastaut Syndrome (LGS). Subjects will be enrolled at approximately 10 investigational sites in the U.S. for up to 15 weeks. Subjects will be randomly assigned to either a low dose or a high dose. The study will include a baseline period, a titration period and a maintenance period. After the maintenance period, subjects will either continue into an open-label extension study or enter the taper period with a final visit 1 week after the last dose.

DETAILED DESCRIPTION:
LGS poses a significant treatment challenge. While antiepileptic medications are the mainstay of treatment, no one antiepileptic drug (AED) provides satisfactory relief for all or most patients with LGS and a combination of treatments is often required. Many patients with LGS are refractory to standard AED treatment.

More effective and better tolerated treatment options are needed for this population of medically intractable epilepsy patients. Clobazam is unique in that it is the only non-1, 4-benzodiazepine used in the treatment of epilepsy.

ELIGIBILITY:
Key Inclusion Criteria:

* Subject must have been <11 years of age at the onset of LGS
* Subject must have LGS
* Subject must be on at least 1 stable dose AED
* Parent or caregiver must be able to keep an accurate seizure diary

Key Exclusion Criteria:

* Etiology of subject's seizures is a progressive neurologic disease. Subjects with tuberous sclerosis will not be excluded from study participation
* Subject has had an episode of status epilepticus within 12 weeks of baseline
* Subject has had an anoxic episode requiring resuscitation within 1 year of screening
* Subject has had a clinically significant history of an allergic reaction or significant sensitivity to benzodiazepines
* Subject is taking more than 3 concurrent AEDs. Note: Vagal Nerve Stimulation (VNS) or ketogenic diet is allowed and each will be counted as one of the three allowed AEDs
* If the subject is on the ketogenic diet, has been for less than 4 weeks prior to screening or suffers from frequent stooling
* If the subject has a VNS, the settings have not been stable for at least 4 weeks prior to screening
* Subject has taken corticotropins in the 6 months prior to screening
* Subject is currently taking long-term systemic steroids (excluding inhaled medication for asthma treatment) or any other daily medication known to exacerbate epilepsy. An exception will be made of prophylactic medication, for example, for urinary tract infections or asthma
* If the subject is taking felbamate, has been taking it for less than 1 year prior to screening or previous treatment with felbamate resulted in withdrawal due to liver or bone marrow adverse events

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (14):
- United States (14):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Pediatric Epilepsy & Neurology Specialists, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Childrens Hospital Boston, Boston, Massachusetts
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - Children's Hospital, Columbus, Ohio
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Dallas Pediatric Neurology Associates, Dallas, Texas
  - Texas Child Neurology, LLP, Plano, Texas
  - Monarch Medical Research, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Conry JA, Ng YT, Paolicchi JM, Kernitsky L, Mitchell WG, Ritter FJ, Collins SD, Tracy K, Kormany WN, Abdulnabi R, Riley B, Stolle J. Clobazam in the treatment of Lennox-Gastaut syndrome. Epilepsia. 2009 May;50(5):1158-66. doi: 10.1111/j.1528-1167.2008.01935.x. Epub 2008 Dec 15. PMID 19170737

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Started | 32 | 36
Completed | 28 | 30
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clobazam Low Dose | Clobazam High Dose | Total
Number analyzed (Participants) | 32 | 36 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30 | 33 | 63
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.18 (5.37) | 8.51 (5.14) | 8.82 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Number of Drop Seizures.
Description: Number of drop seizures (average per week) was obtained from seizure diaries. The average drop in seizures per week for patients who did not complete the maintenance period was calculated based on the time from the beginning of the maintenance period to date of withdrawal.
Time Frame: 4-week baseline period and 4-week maintenance period
Population: Modified Intention-to-Treat (MITT) populations consist of all randomized patients who received study medication and who have both a baseline and post-baseline measurement and have at least one measurement during the maintenance period.
Measure: Mean (Standard Deviation); unit: Percent Reduction
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Number analyzed (Participants) | 29 | 32
Percent Reduction | 10.1 (122.3) | 85.2 (17.1)
Statistical Analysis 1: Comparison: Clobazam Low Dose; Test type: Superiority or Other; p < 0.0182, 1-sided Wilcoxon signed rank test; 1-sided Wilcoxon signed rank test was used to assess the difference from baseline
Statistical Analysis 2: Comparison: Clobazam High Dose; Test type: Superiority or Other; p = 0.0001, 1-sided Wilcoxon signed rank test — 1-sided Wilcoxon signed rank test was used to assess the difference from baseline

2. Secondary Outcome: Percent of Patients Considered Treatment Responders Defined as Those With a >= 25%, >= 50%, >= 75%, and 100% Reduction in Drop Seizures.
Description: as for outcome 1
Time Frame: 4-week baseline period and 4-week maintenance period
Measure: Number; unit: Percent of participants
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Number analyzed (Participants) | 32 | 36
Percent of participants
  ≥ 25% reduction | 18 | 32
  ≥ 50% reduction | 12 | 30
  ≥ 75% reduction | 7 | 23
  100% reduction | 2 | 8

3. Secondary Outcome: Parent/Caregiver Global Evaluations of the Patient's Overall Change in Symptoms.
Description: The parent/caregiver was asked to rate the patient's overall change in symptoms and overall change in seizure activity and Quality of Life since the beginning of clobazam treatment by checking "very much improved", "much improved", "minimally improved", "no change", "minimally worse", "much worse", or "very much worse".
Time Frame: Week 3
Population: MITT population, baseline evaluations compared to Week 3 evaluations.
Measure: Number; unit: participants
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Number analyzed (Participants) | 32 | 36
participants
  Very Much Improved | 7 | 15
  Much Improved | 9 | 15
  Minimally Improved | 9 | 1
  No Change | 3 | 0
  Minimally Worse | 0 | 1
  Much Worse | 1 | 0
  Very Much Worse | 0 | 0

4. Primary Outcome: A Comparison of the High Dose Group to Low Dose Group of the Percent Reduction in Number of Drop Seizures.
Description: as for outcome 1
Time Frame: 4-week baseline period and the 4-week maintenance period
Population: MITT population
Measure: Median (Full Range); unit: Percent Reduction
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Number analyzed (Participants) | 29 | 32
Percent Reduction | 29 [-531 to 100] | 93 [48 to 100]
Statistical Analysis 1: Comparison: Clobazam Low Dose vs Clobazam High Dose; Test type: Non-Inferiority or Equivalence — Assuming a standard deviation of 50%, one-tailed significance at 0.05 and a power of 80% to detect a reduction of at least 25% (baseline to final in a within-subjects design), then approximately 27 subjects would have been required in each treatment arm. Assuming a 10% drop-out rate, then approximately 30 subjects per treatment were to be enrolled in the study; p < 0.0001, 1-sided Wilcoxon Rank-Sum Test; 1-sided Wilcoxon Rank-Sum Test was used to compare the high dose group to the low dose group

5. Secondary Outcome: Parent/Caregiver Global Evaluations of the Patient's Overall Change in Symptoms.
Description: as for outcome 3
Time Frame: Week 7
Population: MITT population, baseline evaluations compared to Week 7 evaluations.
Measure: Number; unit: participants
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Number analyzed (Participants) | 32 | 36
participants
  Very Much Improved | 6 | 16
  Much Improved | 6 | 11
  Minimally Improved | 10 | 1
  No Change | 5 | 0
  Minimally Worse | 1 | 1
  Much Worse | 0 | 0
  Very Much Worse | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 15 weeks
Description: Adverse Events were assessed by the Investigator at the end of the 4 week Baseline period (Day -1) and at weekly/biweekly visits (Weeks 1, 2, 3, 5, 7, 9 and 11) throughout the study.
Arm/Group | Clobazam Low Dose | Clobazam High Dose
Serious Adverse Events (participants affected / at risk) | 1/32 | 3/36
Other Adverse Events (participants affected / at risk) | 27/32 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Clobazam Low Dose (N=32) | Clobazam High Dose (N=36)
Constipation (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sleep Apnea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Clobazam Low Dose (N=32) | Clobazam High Dose (N=36)
Abnormal Behavior (Psychiatric disorders) | 0 | 2
Aggression (Psychiatric disorders) | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Convulsion (Nervous system disorders) | 3 | 1
Coordination abnormal (Nervous system disorders) | 2 | 2
Gastroenteritis viral (Infections and infestations) | 3 | 0
Hypomania (Psychiatric disorders) | 1 | 3
Insomnia (Psychiatric disorders) | 1 | 3
Irritability (General disorders) | 1 | 2
Lethargy (Nervous system disorders) | 3 | 4
Nasopharyngitis (Infections and infestations) | 0 | 4
Otitis media (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pyrexia (General disorders) | 1 | 2
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 3
Sedation (Nervous system disorders) | 2 | 3
Sinusitis (Infections and infestations) | 2 | 2
Skin laceration (Injury, poisoning and procedural complications) | 2 | 2
Somnolence (Nervous system disorders) | 4 | 7
Toothache (Gastrointestinal disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1
Viral infection (Infections and infestations) | 0 | 4
Viral upper respiratory tract infection (Infections and infestations) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Affect lability (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator agrees to delete, at Sponsor's request, from any proposed Public Presentation any information or material that Sponsor deems confidential or proprietary.